CLINICAL TRIAL: NCT01504087
Title: Using Inflammatory Markers to Predict the Development and Outcome of Venous Thromboembolism in an Intensive Care Unit
Brief Title: ICU Venous Thromboembolism Incidence Study in a Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201011022RC
Record Dates: First submitted 2011-07-19; First posted 2012-01-05 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-07

CONDITIONS: Venous Thromboembolism
Keywords: patient in critical care
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patinet with deep venous thrombosis: patient with deep venous thrombosis by ultrasonography as case; patient with no deep venous thrombosis by ultrasonography as control
- patient without deep venous thrombosis

SUMMARY:
Venous thromboembolism (VTE) is one of the major public health problems in Western country. More than 100,000 Americans die each year from VTE. VTE is also a common complication of critical illness,1-2 and probably related to poor outcome in this patient group. Although there are guidelines about VTE prophylaxis in acutely ill medical patients and patients in medical ICU3, they are overlooked in our daily practice frequently in our country. There are many reasons for our common practice, including inadequate knowledge for the ICU physicians, more patients with bleeding tendency in ICU and low prevalence of VTE in our (eastern) country. However, the true prevalence of VTE in ICU and if thromboprophylaxis still needed in certain high risk patients are not unknown. Besides, if there is a difference in the VTE rate between western and eastern patients, what is the underlying mechanism? The major objective of this application is to answer the first part of the problem, i.e. to delineate the scope of this problem.

The specific aims of this application are as follows:

* prevalence of venous thromboembolism in ICU in Taiwan
* specific risk in subgroups of ICU patients
* prevalence and risk factors for silent pulmonary embolism

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to medical ICU with age over 18 y/o are eligible

Exclusion Criteria:

* Patients who do not sign the informed consent will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to ICU with age over 18 y/o are eligible
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-05

PRIMARY OUTCOMES:
deep venous thrombosis by ultrasound | day 14 after ICU admission

SECONDARY OUTCOMES:
any clinical thromboembolic event | day 14

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Wei Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Yunlin branch, Douliu, Taiwan, Taiwan